CLINICAL TRIAL: NCT02532829
Title: Effects of Different Metabolic States and Surgical Models on Glucose Metabolism and Secretion of Ileal L-cell Peptides
Brief Title: Human Intestinal Peptides Evaluation and Research
Acronym: HIPER
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Turkish Metabolic Surgery Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/H01
Record Dates: First submitted 2015-08-13; First posted 2015-08-26 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- GROUP NS-A: Healthy Participants: No known disease, no previous surgery, HbA1c<5.7%, BMI<25 kg/m2 (n=30). Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- GROUP NS-B: Obese, type 2 diabetic: Type 2 diabetes diagnosis longer than 3 years; BMI>30 kg/m2 (n=30). Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- GROUP NS-C: Non-obese, type 2 diabetic: Type 2 diabetes diagnosis longer than 3 years; BMI<30 kg/m2 (n=30). Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- GROUP NS-D: Obese non-diabetic: HbA1c<5.7%, No signs and history of T2D, and BMI>30 kg/m2 (n=30). Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- Group SG: Type 2 Diabetic participants who underwent a sleeve gastrectomy, performed more than 6 months ago, but within the last 2 years, with steady weight profile. Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- Group MGB: Type 2 Diabetic participants who underwent a mini-gastric bypass, performed more than 6 months ago, but within the last 2 years, with steady weight profile. Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- Group IT: Type 2 Diabetic participants who underwent a sleeve gastrectomy with ileal transposition, performed more than 6 months ago, but within the last 2 years, with steady weight profile. Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis
- Group TB: Type 2 Diabetic participants who underwent a sleeve gastrectomy with transit bipartition, performed more than 6 months ago, but within the last 2 years, with steady weight profile. Blood sample analysis (Blood samples will be taken for the analysis of GLP-1, Peptide YY, glucose and insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test).
  Interventions: Other: blood sample analysis

INTERVENTIONS:
Other: blood sample analysis — Measurement of GLP-1, Peptide YY, Glucose and Insulin before and 30-60-120 minutes after Oral Mixed Meal Tolerance Test.

SUMMARY:
The HIPER-1 study is a single centre cross sectional study in which a total of 240 participants (in different metabolic states and surgical models) will receive an Oral Mixed Meal Tolerance Test (OMTT). At baseline and after 30, 60 and 120 minutes the PYY levels, GLP-1 levels, glucose and insulin sensitivity will be measured. The primary endpoint of the study will be the area under the GLP-1 and Peptide - YY curves and insulin sensitivity following the OMTT.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes mellitus (T2DM) are increasing worldwide, thus reaching pandemic proportions. Diet, exercise and medication remain the cornerstones of type 2 diabetes mellitus treatment. But, apart from studies demonstrating promising results in some of the developed countries; the long-term success rates of lifestyle and drug modifications are disappointing. In cases where classic strategies proved to be inadequate, broad type of gastrointestinal (GI) surgery methods offer new alternatives to treat obesity and T2DM. The variable levels of incretin stimulation (especially GLP-1) and improved glycaemic control in those with diabetes have been shown following various bariatric techniques.

Therefore, investigators aimed to analyze the levels of GLP-1 and Peptide YY hormones together with indices of insulin sensitivity in participants with various health conditions and in participants who underwent different surgical options including sleeve gastrectomy, minigastric bypass, sleeve gastrectomy with ileal transposition and sleeve gastrectomy with transit bipartition.

ELIGIBILITY:
For NON-SURGERY GROUPS

Inclusion Criteria:

1. GROUP NS-A: Healthy participants, no known disease, no previous surgery, HbA1c<5.7%, BMI<25 kg/m2 (n=30).

   GROUP NS-B: Obese diabetic, type 2 diabetes diagnosis longer than 3 years; BMI>30 kg/m2 (n=30).

   GROUP NS-C: Non-obese diabetic, type 2 diabetes diagnosis longer than 3 years; BMI<30 kg/m2 (n=30).

   GROUP NS-D: Obese non-diabetics, HbA1c<5.7%, No signs and history of T2D, and BMI>30 kg/m2 (n=30).
2. Preferably not on any kind of anti-diabetic drugs or will accept cessation of all anti-diabetic drugs 2 days prior to evaluation.
3. Absence of co-morbidities (dyslipidemia, hypertension, neuropathy, retinopathy, cardiovascular disease, stroke events or lower extremity amputation).
4. Possibility to participate to the quadruplicate measurement protocol.

Exclusion Criteria:

1. Anti insulin / islet antibody and glutamic acid decarboxylase antibody (antiGAD) positivity, plasma fasting C-peptide lesser than 1 ng/ml.
2. Liver cirrhosis, severe renal failure, collagen diseases, severe endocrinopathies, blindness.
3. Heart failure, acute myocardial infarction, stroke or transient ischemic attack, unstable angina pectoris.
4. History of malignancy or malignant neoplasm in place, severe inflammatory complications, neurological or cardiovascular in act.
5. Pregnancy
6. Any conditions that at the discretion of the head of the study can represent risk to the participant or could affect the protocol results.

For SURGERY GROUPS

Inclusion Criteria:

1. Type 2 Diabetic participants who underwent a sleeve gastrectomy, a mini-gastric bypass, a sleeve gastrectomy with ileal transposition or a sleeve gastrectomy with transit bipartition performed more than 6 months ago, but within the last 2 years, with steady weight profile.
2. Preferably not on any kind of anti-diabetic drugs or will accept cessation of all anti-diabetic drugs 2 days prior to evaluation.
3. Absence of or resolved co-morbidities (dyslipidemia, hypertension, neuropathy, retinopathy, cardiovascular disease, stroke events or lower extremity amputation).
4. Possibility to participate to the quadruplicate measurement protocol.

Exclusion Criteria:

1. Liver cirrhosis, severe renal failure, collagen diseases, severe endocrinopathies, blindness.
2. Heart failure, acute myocardial infarction, stroke or transient ischemic attack, unstable angina pectoris.
3. History of malignancy or malignant neoplasm in place, severe inflammatory complications, neurological or cardiovascular in act.
4. Pregnancy
5. Any conditions that at the discretion of the head of the study can represent risk to the participant or could affect the protocol results.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. GROUP NS-A: Healthy participants, no known disease, no previous surgery, HbA1c<5.7%, BMI<25 kg/m2.
  2. GROUP NS-B: Obese diabetic, type 2 diabetes diagnosis longer than 3 years; BMI>30 kg/m2.
  3. GROUP NS-C: Non-obese diabetic, type 2 diabetes diagnosis longer than 3 years; BMI<30 kg/m2.
  4. GROUP NS-D: Obese non-diabetics, HbA1c<5.7%, No signs and history of T2D, and BMI>30 kg/m2.
  5. Group SG: Participants who underwent sleeve gastrectomy
  6. Group MGB: Participants who underwent mini-gastric bypass
  7. Group IT: Participants who underwent sleeve gastrectomy with ileal transposition
  8. Group TB: Participants who underwent sleeve gastrectomy with transit bipartition
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Plasma GLP-1 and P-YY measurements by ELISA in participants with various health conditions. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test and results will be expressed as pmol/L.
Plasma GLP-1 and P-YY measurements by ELISA in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test and results will be expressed as pmol/L.

SECONDARY OUTCOMES:
Body Mass Index (BMI) in participants with various health conditions. | Up to 6 months.
  BMI will be expressed in kg/m^2 (weight in kilograms and height in meters).
Body Mass Index (BMI) in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  BMI will be expressed in kg/m^2 (weight in kilograms and height in meters).
Waist and hip circumference in participants with various health conditions. | Up to 6 months.
  Waist and hip circumferences will be expressed as centimeters.
Waist and hip circumference in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Waist and hip circumferences will be expressed as centimeters.
Plasma glucose levels in participants with various health conditions. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test. Plasma glucose levels will be measured by Enzymatic Hexokinase method and results will be expressed as mg/dl.
Plasma glucose levels in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test. Plasma glucose levels will be measured by Enzymatic Hexokinase method and results will be expressed as mg/dl.
Plasma insulin levels in participants with various health conditions. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test. Plasma insulin levels will be measured by ECLIA method and results will be expressed as mU/ml.
Plasma insulin levels in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Measurements will be performed before and 30-60-120 minutes after a mixed meal test. Plasma insulin levels will be measured by ECLIA method and results will be expressed as mU/ml.

OTHER OUTCOMES:
Plasma HbA1c levels in participants with various health conditions. | Up to 6 months.
  Measurements will be performed in the fasting state using the Turbidometric Assay and results will be expressed as percentage (%).
Plasma HbA1c levels in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Measurements will be performed in the fasting state using the Turbidometric Assay and results will be expressed as percentage (%).
Plasma Liver Function Tests (SGOT, SGPT and GGT levels) in participants with various health conditions. | Up to 6 months.
  Measurements will be performed in the fasting state using IFCC Enzymatic Assay and results will be expressed as U/L.
Plasma Liver Function Tests (SGOT, SGPT and GGT levels) in participants treated by different bariatric and metabolic surgical techniques. | Up to 6 months.
  Measurements will be performed in the fasting state using IFCC Enzymatic Assay and results will be expressed as U/L.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Celik, MD, Study Director — Turkish Metabolic Surgery Foundation

REFERENCES:
- [Result] DePaula AL, Macedo AL, Schraibman V, Mota BR, Vencio S. Hormonal evaluation following laparoscopic treatment of type 2 diabetes mellitus patients with BMI 20-34. Surg Endosc. 2009 Aug;23(8):1724-32. doi: 10.1007/s00464-008-0168-6. Epub 2008 Oct 2. PMID 18830747
- [Result] Kashyap SR, Daud S, Kelly KR, Gastaldelli A, Win H, Brethauer S, Kirwan JP, Schauer PR. Acute effects of gastric bypass versus gastric restrictive surgery on beta-cell function and insulinotropic hormones in severely obese patients with type 2 diabetes. Int J Obes (Lond). 2010 Mar;34(3):462-71. doi: 10.1038/ijo.2009.254. Epub 2009 Dec 22. PMID 20029383
- [Result] Finelli C, Padula MC, Martelli G, Tarantino G. Could the improvement of obesity-related co-morbidities depend on modified gut hormones secretion? World J Gastroenterol. 2014 Nov 28;20(44):16649-64. doi: 10.3748/wjg.v20.i44.16649. PMID 25469034
- [Result] Goldfine AB, Mun EC, Devine E, Bernier R, Baz-Hecht M, Jones DB, Schneider BE, Holst JJ, Patti ME. Patients with neuroglycopenia after gastric bypass surgery have exaggerated incretin and insulin secretory responses to a mixed meal. J Clin Endocrinol Metab. 2007 Dec;92(12):4678-85. doi: 10.1210/jc.2007-0918. Epub 2007 Sep 25. PMID 17895322
- [Result] Kashyap SR, Bhatt DL, Wolski K, Watanabe RM, Abdul-Ghani M, Abood B, Pothier CE, Brethauer S, Nissen S, Gupta M, Kirwan JP, Schauer PR. Metabolic effects of bariatric surgery in patients with moderate obesity and type 2 diabetes: analysis of a randomized control trial comparing surgery with intensive medical treatment. Diabetes Care. 2013 Aug;36(8):2175-82. doi: 10.2337/dc12-1596. Epub 2013 Feb 25. PMID 23439632
- [Result] Troke RC, Tan TM, Bloom SR. The future role of gut hormones in the treatment of obesity. Ther Adv Chronic Dis. 2014 Jan;5(1):4-14. doi: 10.1177/2040622313506730. PMID 24381724
- [Result] Essah PA, Levy JR, Sistrun SN, Kelly SM, Nestler JE. Effect of weight loss by a low-fat diet and a low-carbohydrate diet on peptide YY levels. Int J Obes (Lond). 2010 Aug;34(8):1239-42. doi: 10.1038/ijo.2010.48. Epub 2010 Mar 30. PMID 20351741
- [Result] Batterham RL, Cohen MA, Ellis SM, Le Roux CW, Withers DJ, Frost GS, Ghatei MA, Bloom SR. Inhibition of food intake in obese subjects by peptide YY3-36. N Engl J Med. 2003 Sep 4;349(10):941-8. doi: 10.1056/NEJMoa030204. PMID 12954742
- [Result] Santoro S. From Bariatric to Pure Metabolic Surgery: New Concepts on the Rise. Ann Surg. 2015 Aug;262(2):e79-80. doi: 10.1097/SLA.0000000000000590. No abstract available. PMID 24646534
- [Result] Celik A, Ugale S. Functional restriction and a new balance between proximal and distal gut: the tools of the real metabolic surgery. Obes Surg. 2014 Oct;24(10):1742-3. doi: 10.1007/s11695-014-1368-x. No abstract available. PMID 25027983
- [Derived] Cagiltay E, Celik A, Dixon JB, Pouwels S, Santoro S, Gupta A, Ugale S, Abdul-Ghani M. Effects of different metabolic states and surgical models on glucose metabolism and secretion of ileal L-cell peptides: results from the HIPER-1 study. Diabet Med. 2020 Apr;37(4):697-704. doi: 10.1111/dme.14191. Epub 2019 Dec 15. PMID 31773794
- [Derived] Celik A, Dixon JB, Pouwels S, Celik BO, Karaca FC, Gupta A, Santoro S, Ugale S. Effects of different metabolic states and surgical models on glucose metabolism and secretion of ileal L-cell peptides: protocol for a cross-sectional study. BMJ Open. 2016 Mar 14;6(3):e010245. doi: 10.1136/bmjopen-2015-010245. PMID 26975937